CLINICAL TRIAL: NCT03234309
Title: High Resolution Steady State Blood Volume Maps in Pediatric Brain Tumors Using MRI
Brief Title: Ferumoxytol in Magnetic Resonance Imaging of Pediatric Patients With Brain Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No enrollments
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00016165; NCI-2017-00713 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016165 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Ferrosoferric Oxide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (ferumoxytol, MRI) (Experimental): Patients undergo MRI with GBCA per standard of care over 45-60 minutes and then receive ferumoxytol IV followed by MRI over 10 minutes on day 1. Patients may optionally undergo MRI over 30 minutes without any contrast agent on day 2. Each study visit consisting of 2 days may repeat no more frequently than 4 weeks for up to 5 study visits at different stages of the disease as determined by the investigator.
  Interventions: Drug: Ferumoxytol; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Ferumoxytol — Given IV
  Other Names: Feraheme; Ferumoxytol Non-Stoichiometric Magnetite
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This phase II trial studies ferumoxytol in the magnetic resonance imaging of pediatric patients with brain tumors. Magnetic resonance imaging using ferumoxytol may help in viewing a brain tumor and blood vessels in and around the tumor in a different way than the standard gadolinium-based contrast agent. Imaging with this experimental contrast agent may give doctors more information about tumor blood supply and the extent of the tumor itself.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Testing the superiority of ferumoxytol-based steady state (SS)-cerebral blood volume (CBV) maps over gadolinium-based contrast agent (GBCA)-based dynamic susceptibility weighted (DSC)-CBV maps in visualizing pediatric brain tumor blood volume maps.

SECONDARY OBJECTIVES:

I. Correlation of relative cerebral blood volume (rCBV) with histology and genetic markers.

II. Assessment of therapeutic response. III. Assessment of late ferumoxytol enhancement at various stages of disease.

OUTLINE:

Patients undergo magnetic resonance imaging (MRI) with GBCA per standard of care over 45-60 minutes and then receive ferumoxytol intravenously (IV) followed by MRI over 10 minutes on day 1. Patients may optionally undergo MRI over 30 minutes without any contrast agent on day 2. Each study visit consisting of 2 days may repeat no more frequently than 4 weeks for up to 5 study visits at different stages of the disease as determined by the investigator.

After completion of study, patients are followed up at 2 and 6 weeks and then periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a presumed diagnosis of brain tumor (based on imaging) or a confirmed brain tumor (based on pathology) before or after any oncologic treatment (surgery/chemotherapy/radiation)
* All subjects, or their legal guardians, must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines
* Subjects with a calculated glomerular filtration rate (GFR) > 60 mL/min/1.73 m^2
* Sexually active women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; surgical intervention i.e. tubal ligation or vasectomy; post-menopausal > 6 months or abstinence) for at least two months after each cycle of the study; should a female become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Subjects with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible
* Subjects with known allergic or hypersensitivity reactions to parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations (Ferumoxytol Investigator's Drug Brochure, 2009); subjects with significant drug or other allergies or autoimmune diseases may be enrolled at the investigator's discretion
* Subjects who are pregnant or lactating or who suspect they might be pregnant
* Subjects who have a contraindication for 3Tesla (3T) MRI: metal in their bodies (a cardiac pacemaker or other incompatible device), are severely agitated, or have an allergy to gadolinium containing contrast material
* Subjects with known iron overload (genetic hemochromatosis); in subjects with a family history of hemochromatosis, hemochromatosis must be ruled out prior to study entry with normal values of the following blood tests: transferrin saturation (TS) test and serum ferritin (SF) test; all associated costs will be paid by the study
* Subject who have received ferumoxytol within 4 weeks of study entry

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Overlay accuracy with 3-dimensional anatomical T1w post contrast scans | Up to 5 years
  Ferumoxytol-based steady state-cerebral blood volume maps will be compared to gadolinium-based dynamic susceptibility weighted-cerebral blood volume maps using a 3-point scale. The mean score between the two readers will be used in the primary analyses. Inter-reader agreement will be assessed using weighted Kappa to make sure that the visualization variables are used reliably.
Confidence in identifying the lesion corresponding areas on cerebral blood volume maps | Up to 5 years
  The mean score between the two readers will be used in the primary analyses. A linear mixed effects model will be used to compare the mean of the four visualization variables between steady state and dynamic susceptibility weighted overall and at each of time points while taking into account the correlation due to repeated measures within the same patient. Inter-reader agreement will be assessed using weighted Kappa to make sure that the visualization variables are used reliably.
Cerebral blood volume in small (< 1 cm) enhancing lesions | Up to 5 years
  Ferumoxytol-based steady state-cerebral blood volume maps will be compared to gadolinium-based dynamic susceptibility weighted-cerebral blood volume maps using a 3-point scale.
Delineation of tumor from larger blood vessels | Up to 5 years
  Ferumoxytol-based steady state-cerebral blood volume maps will be compared to gadolinium-based dynamic susceptibility weighted-cerebral blood volume maps using a 3-point scale. The mean score between the two readers will be used in the primary analyses. Inter-reader agreement will be assessed using weighted Kappa to make sure that the visualization variables are used reliably.

SECONDARY OUTCOMES:
Relative cerebral blood volume value | Up to 5 years
  Sensitivity and specificity of relative cerebral blood volume will be calculated for identifying true disease progression at different cutoff points and compare the performance between steady state and dynamic susceptibility weighted maps using McNemar's tests, and using a mixed effect logistic regression model to look at all data across different disease stages (within the same patient) if necessary and allowed by available data.
Treatment response | Up to 5 years
  For the assessment of therapeutic response, enhancing areas will be categorized as active tumor or therapy related changes based on relative cerebral blood volume values. Different cutoff points (e.g. 1.5, 1.75 and 2) will be tested for relative cerebral blood volume value from both steady state and dynamic susceptibility weighted maps, and disease status will be confirmed with subsequent magnetic resonance imaging results as recommended by Response Assessment in Neuro-Oncology Criteria or histopathology from additional surgeries ("gold standard").
Histology and genetic markers | Up to 5 years
  A linear model will be used to assess correlation of relative cerebral blood volume with histology and genetic markers based on the availability of data and type of tumor.
Ferumoxytol enhancement | At 24 hours after administration
  Similar models to those for primary objectives will evaluate late ferumoxytol enhancement at various stages of disease. Will be assessed on T1 and T2 weighted magnetic resonance (MR) sequences. Enhancement changes including intensity and pattern (heterogeneity) at various stages of disease will be analyzed and compared to gadolinium based contrast agent (GBCA).
Survival | Up to 5 years
  Data will be collected for 5 years.
Progression free survival | Up to 5 years
  Data will be collected for 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, Principal Investigator — OHSU Knight Cancer Institute